CLINICAL TRIAL: NCT07137624
Title: Effects of Motor Imagery and Action Observation on Gait Initiation and Spatiotemporal Gait Parameters in Multiple Sclerosis
Brief Title: Motor Imagery and Action Observation for Gait Function in MS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Merve Ünal, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FTREK25/48
Record Dates: First submitted 2025-08-06; First posted 2025-08-22 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis
Keywords: Motor imagery; Action Observation
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the experimental group (motor imagery + action observation) or the control group (nature video).
Who Masked: Participant
Masking Description: The study will be single-blinded. Participants will not be informed of their group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Arm 1: Experimental Group: Action Observation + Motor Imagery
  Interventions: Behavioral: Action Observation + Motor Imagery
- Arm 2 (Other): Arm 2: Control Group: Nature video
  Interventions: Behavioral: Nature Video

INTERVENTIONS:
Behavioral: Action Observation + Motor Imagery — Participants will watch videos showing walking actions and will be instructed to mentally simulate the movement.
  Arms: Arm 1
Behavioral: Nature Video — Participants will watch a video of nature scenes.
  Arms: Arm 2

SUMMARY:
This study will investigate whether mentally simulating walking movements while watching others walk can improve walking performance in individuals with Multiple Sclerosis (MS). Participants will be divided into two groups: one group will watch walking videos and imagine themselves walking, while the other group will watch nature scenes. The study will measure muscle activity and walking patterns to assess the effects. The results may help support the use of mental practice techniques to improve mobility in people with MS.

DETAILED DESCRIPTION:
This study aims to explore the impact of mental simulation of walking movements on walking performance in individuals with Multiple Sclerosis (MS). The participants will be randomly assigned to two groups: the experimental group will watch walking-related videos and engage in mental imagery exercises, imagining themselves walking, while the control group will watch nature scenes without any walking-related content.

Objectives:

To determine whether mental imagery can enhance walking ability and gait parameters in individuals with MS.

To measure the effect of mental simulation on muscle activity and walking patterns, including stride length, walking speed, and balance.

Study Procedure:

The study will consist of multiple sessions, where participants will first undergo baseline assessments of walking ability. Following this, they will engage in either the walking video and imagery task (experimental group) or the nature video viewing task (control group) for a predetermined period of time. Measurements of muscle activity using electromyography (EMG) and walking patterns will be recorded before and after the intervention.

Potential Impact:

The results from this study may provide insights into the use of mental practice techniques as a non-invasive intervention to improve mobility in individuals with MS, a population often affected by walking difficulties. Mental imagery could serve as an adjunct therapy to traditional physical rehabilitation methods.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of multiple sclerosis (MS) by a neurologist
* No history of relapse within the past 3 months and not currently experiencing a relapse
* A score of 24 or higher on the standardized Mini Mental State Examination

Exclusion Criteria:

* Presence of serious health conditions affecting the muscles, heart, lungs, or metabolism that could interfere with participation
* History of other neurological disorders, head injury, or chronic psychiatric conditions
* Chronic pain lasting longer than six months
* Significant muscle stiffness in the legs that may affect EMG recordings
* Hearing difficulties
* Vision problems as determined by the Snellen visual acuity test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Change in Tibialis Anterior and Gastrocnemius Medialis Muscle Activity Amplitude | Before and immediately after the intervention
  Change in muscle activity amplitude (microvolts, µV) of tibialis anterior and gastrocnemius medialis during gait initiation measured by surface EMG.
Change in Tibialis Anterior and Gastrocnemius Medialis Muscle Activity Onset Latency | Before and immediately after the intervention.
  Change in onset latency (milliseconds, ms) of tibialis anterior and gastrocnemius medialis muscle activation during gait initiation measured by surface EMG.
Change in Step Length | Before and immediately after the intervention
  Change in step length (centimeters, cm) during gait initiation measured by the GAITRite system.
Change in Step Time | Before and immediately after the intervention
  Change in step time (seconds, s) during gait initiation measured by the GAITRite system.
Change in Step Width | Before and immediately after the intervention
  Change in step width (centimeters, cm) during gait initiation measured by the GAITRite system.
Change in Double Support Period | Before and immediately after the intervention
  Change in double support period (percentage of gait cycle, %) during gait initiation measured by the GAITRite system.
Change in Gait Velocity | Before and immediately after the intervention
  Change in gait velocity (centimeters per second, cm/s) during gait initiation measured by the GAITRite system.
Change in Cadence | Before and immediately after the intervention
  Change in cadence (steps per minute, steps/min) during gait initiation measured by the GAITRite system.

SECONDARY OUTCOMES:
Motor Imagery Vividness | Baseline only
  Kinesthetic and visual imagery vividness will be assessed using the Kinesthetic and Visual Imagery Questionnaire-20 (KVIQ-20), which includes 10 visual and 10 kinesthetic items (20 total). Each item is rated on a 5-point Likert scale (1 = no image/sensation, 5 = vivid image/sensation). Higher scores indicate better imagery ability.
Mental Chronometry Ratio | Baseline only
  The ratio between imagined and actual Timed Up and Go (TUG) performance time (both measured in seconds, s) will be calculated. During imagined trials, participants will press a button to mark the start and end of the imagined movement sequence. A ratio closer to 1 indicates better temporal congruence between imagined (iTUG) and executed TUG performance.
Limb Laterality Recognition Performance | Baseline only
  Right-left discrimination ability will be evaluated using the Recognise Foot App™ developed by the NOI Group™. Both accuracy (percentage of correct responses, %) and response time (milliseconds, ms) will be recorded.
Cognitive Status | Baseline only
  General cognitive functioning will be screened using the Standardized Mini-Mental State Examination (SMMSE). The test is scored on a 30-point scale (0-30). Scores ≥24 indicate normal cognitive functioning.
Fatigue Level | Baseline only
  Fatigue severity specific to MS will be measured with the Fatigue Severity Scale (FSS). The FSS consists of 9 items rated on a 7-point Likert scale (1 = strongly disagree; 7 = strongly agree). The final score is calculated as the mean of all items (range: 1-7), with higher scores indicating greater fatigue severity.
Anxiety and Depression | Baseline only
  Emotional state will be assessed using the Hospital Anxiety and Depression Scale (HADS). The scale consists of 14 items divided into two subscales: anxiety (7 items) and depression (7 items). Each item is scored from 0 to 3, yielding subscale scores ranging from 0 to 21. Higher scores indicate greater levels of anxiety or depression.
Disability Level | Baseline only
  Expanded Disability Status Scale (EDSS) scoring will be performed using the standardized Neurostatus-EDSS format. This scale evaluates functional systems such as motor ability, balance, vision, and sensory function to quantify disability level in individuals with multiple sclerosis. Scores range from 0 to 10 in 0.5-point increments, where 0 indicates normal neurological status and 10 represents death due to MS. Higher scores reflect greater disability.
Visual Acuity | Baseline only
  Participants' visual acuity will be assessed using the Snellen chart under standard conditions. The test will be conducted with or without corrective lenses depending on the participant's usual visual aid usage. Visual acuity will be recorded as a Snellen fraction (e.g., 20/20, 20/40), where larger denominators indicate poorer visual performance.

OTHER OUTCOMES:
Perceived Task Load | Immediately after the intervention
  The NASA Task Load Index (NASA-TLX) will be used to measure mental and physical workload related to the task. The scale consists of six subscales: mental demand, physical demand, temporal demand, performance, effort, and frustration. Each subscale is rated on a 0-100 visual analog scale, and an overall workload score is obtained by averaging the six subscales. Higher scores indicate greater perceived workload.

CONTACTS AND LOCATIONS:
Overall Officials: Yeliz Salcı, Assoc. Prof., Study Chair — Hacettepe University
Locations (1):
- Hacettepe University, Faculty of Physical Therapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wright DJ, Williams J, Holmes PS. Combined action observation and imagery facilitates corticospinal excitability. Front Hum Neurosci. 2014 Nov 27;8:951. doi: 10.3389/fnhum.2014.00951. eCollection 2014. PMID 25505880
- [Background] Rocca MA, Meani A, Fumagalli S, Pagani E, Gatti R, Martinelli-Boneschi F, Esposito F, Preziosa P, Cordani C, Comi G, Filippi M. Functional and structural plasticity following action observation training in multiple sclerosis. Mult Scler. 2019 Oct;25(11):1472-1487. doi: 10.1177/1352458518792771. Epub 2018 Aug 7. PMID 30084706
- [Background] Gil-Bermejo-Bernardez-Zerpa A, Moral-Munoz JA, Lucena-Anton D, Luque-Moreno C. Effectiveness of Motor Imagery on Motor Recovery in Patients with Multiple Sclerosis: Systematic Review. Int J Environ Res Public Health. 2021 Jan 9;18(2):498. doi: 10.3390/ijerph18020498. PMID 33435410
- [Background] Chye S, Valappil AC, Wright DJ, Frank C, Shearer DA, Tyler CJ, Diss CE, Mian OS, Tillin NA, Bruton AM. The effects of combined action observation and motor imagery on corticospinal excitability and movement outcomes: Two meta-analyses. Neurosci Biobehav Rev. 2022 Dec;143:104911. doi: 10.1016/j.neubiorev.2022.104911. Epub 2022 Nov 5. PMID 36349570
- [Background] Salamci M, Salci Y, Topuz S, Yalcin AI, Acar Ozen P, Tuncer A. Gait initiation in multiple sclerosis patients with and without functional loss. Mult Scler Relat Disord. 2023 Nov;79:104990. doi: 10.1016/j.msard.2023.104990. Epub 2023 Sep 4. PMID 37708821